CLINICAL TRIAL: NCT05383638
Title: Effectiveness of Health Promotion Interventions in Improving Patient Satisfaction With Primary Health Services
Brief Title: Effectiveness of Health Promotion Interventions in Improving Patient Satisfaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Li Huan, Doctoral candidate, Universiti Tunku Abdul Rahman
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Drweijie
Record Dates: First submitted 2022-03-16; First posted 2022-05-20 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Primary Health Care; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health promotion (Other): Health education and popularization of science
  Interventions: Other: Health education

INTERVENTIONS:
Other: Health education — Intervention is achieved through health education. Analyze the factors that may affect patients' satisfaction with primary medical services through existing data, and carry out targeted health education.

SUMMARY:
This study investigated whether health promotion intervention can effectively affect patients' satisfaction with primary health care services through questionnaire survey.

DETAILED DESCRIPTION:
The world Health Organization in the 21st century Health Strategy plans new Vision for Human Health and Health Promotion proposed that the main way to maintain human health in the 21st century is health education. Health promotion is an important part of primary health care and the preferred strategy to solve public health problems. Evaluation of patient satisfaction is a key determinant of medical quality and has become an important issue in the evaluation of medical system. The purpose of this study was to explore the effectiveness of health promotion intervention in improving patients' satisfaction with primary health services, explore effective measures for improving patient satisfaction in different regions, and promote the rapid and balanced development of primary health services.

Design：Due to the large difference in economic conditions among different regions of Xi 'this study is divided into two parts:

Phase I: investigation in the main urban area of Xi 'an, understanding the current status of primary health services in the main urban area, and exploring the impact of health promotion on patient satisfaction.

Using Multi stage sampling, 1. Simple random method (clinic), 12 were selected from all primary health care institutions in the main urban area of Xi 'an. 2. Systematic random sampling (patients). Of the 12 institutions sampled, A systematic allocation was used to choose patient based on their registration number. Patients with odds number were assigned to the intervention group, even number was assigned to the control group using the flip coin method. Patients in the intervention group received health promotion interventions, while patients in the control group only received daily greetings. The patients' satisfaction was assessed before and after the intervention and the effectiveness of the intervention was discussed.

Phase II: Research the economically underdeveloped areas outside the main urban area of Xi 'an.

The experience of Phase I was analyzed, intervention measures were improved, an appropriate sample size was selected with the same method as in the first phase, social demographic characteristics of patients and patient satisfaction were measured before and after the investigation, the satisfaction status of patients outside the main urban area of Xi 'an on primary health services was learned, and effective intervention measures were summarized. Finally, to promote the optimal allocation of medical resources in Xi 'an and improve the fairness and accessibility of primary medical services in Xi 'an.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Being able to read and write in Chinese
* Owning a smartphone and knowing how to use WeChat
* Clear consciousness, can communicate normally, can understand the questionnaire correctly.

Exclusion Criteria:

·Patients with mental disorders, cognitive impairment, severe and terminal illness were unable to cooperate with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction after the intervention by using PSQ 18 questionnaires | 6 months
  When contacting the patient for the first time, add the patient's WeChat account and ask the patient to follow the health intervention subscription number. The patient who follows the subscription account can read the intervention materials and watch the intervention videos anytime and anywhere and can also leave the comments and questions. They will also be encouraged to check the text messages and messages previously sent through WeChat subscription accounts, interact with investigators individually through WeChat personal information platform, and discuss with other patients in WeChat groups Participants can seek help through WeChat personal information platform or by phone at any time. We release at least one health intervention data every week, and contact the people being interfered to ensure that the intervention is effective.

CONTACTS AND LOCATIONS:
Overall Officials: MON MIN SWE KYE, DR, Principal Investigator — Tunku Abdul Rahman University
Locations (1):
- Xi 'an Medical University, Xi’an, Shanxi, China